CLINICAL TRIAL: NCT03254940
Title: Charge: Optimizing a Standalone Text Messaging-Based Weight Loss Intervention
Brief Title: Charge: A Text Messaging-based Weight Loss Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: D0752
Record Dates: First submitted 2017-07-12; First posted 2017-08-21 (Actual); Results first posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Weight Loss; Obesity
Keywords: text message; digital health; weight loss; personalized
MeSH Terms: conditions — Weight Loss; Obesity | interventions — Fees and Charges

STUDY DESIGN:
Intervention Model Description: The investigators will use a full factorial design to randomize participants to experimental conditions that reflect the texting intervention components: motivational messaging (self- vs expert-generated), texting frequency (daily vs weekly), reminders (one reminder v. multiple reminders), feedback type (summary score v. specific feedback) and comparison unit (to self v. to a group of people). The full factorial design is power efficient, logistically feasible (because we manipulate conditions using technology) and will allow the investigators to examine the most important main and interaction effects among components.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (32):
- Arm 1: WT-SM-OR-SS-CS (Experimental): Charge: weekly tracking, self-generated motivational messages, one reminder, summary score, compare to self
  Interventions: Behavioral: Charge
- Arm 2: WT-SM-OR-SS-CG (Experimental): Charge: weekly tracking, self-generated motivational messages, one reminder, summary score, compare to group
  Interventions: Behavioral: Charge
- Arm 3: WT-SM-OR-SF-CS (Experimental): Charge: weekly tracking, self-generated motivational messages, one reminder, specific goal feedback, compare to self
  Interventions: Behavioral: Charge
- Arm 4: WT-SM-OR-SF-CG (Experimental): Charge: weekly tracking, self-generated motivational messages, one reminder, specific goal feedback, compare to group
  Interventions: Behavioral: Charge
- Arm 5: WT-SM-MR-SS-CS (Experimental): Charge: weekly tracking, self-generated motivational messages, multiple reminders, summary score, compare to self.
  Interventions: Behavioral: Charge
- Arm 6: WT-SM-MR-SS-CG (Experimental): Charge: weekly tracking, self-generated motivational messages, multiple reminders, summary score, compare to group.
  Interventions: Behavioral: Charge
- Arm 7: WT-SM-MR-SF-CS (Experimental): Charge: weekly tracking, self-generated motivational messages, multiple reminders, specific feedback, compare to self
  Interventions: Behavioral: Charge
- Arm 8: WT-SM-MR-SF-CG (Experimental): Charge: weekly tracking, self-generated motivational messages, multiple reminders, specific feedback, compare to group
  Interventions: Behavioral: Charge
- Arm 9: WT-EM-OR-SS-CS (Experimental): Charge: weekly tracking, expert-generated motivational messages, one reminder, summary score, compare to self
  Interventions: Behavioral: Charge
- Arm 10: WT-EM-OR-SS-CG (Experimental): Charge: weekly tracking, expert-generated motivational messages, one reminder, summary score, compare to group
  Interventions: Behavioral: Charge
- Arm 11: WT-EM-OR-SF-CS (Experimental): Charge: weekly tracking, expert-generated motivational messages, one reminder, specific goal feedback, compare to self
  Interventions: Behavioral: Charge
- Arm 12: WT-EM-OR-SF-CG (Experimental): Charge: weekly tracking, expert-generated motivational messages, one reminder, specific goal feedback, compare to group.
  Interventions: Behavioral: Charge
- Arm 13: WT-EM-MR-SS-CS (Experimental): Charge: weekly tracking, expert-generated motivational messages, multiple reminders, summary score, compare to self
  Interventions: Behavioral: Charge
- Arm 14: WT-EM-MR-SS-CG (Experimental): Charge: weekly tracking, expert-generated motivational messages, multiple reminders,summary score, compare to group
  Interventions: Behavioral: Charge
- Arm 15: WT-EM-MR-SF-CS (Experimental): Charge: weekly tracking, expert-generated motivational messages, multiple reminders, specific goal feedback, compare to self
  Interventions: Behavioral: Charge
- Arm 16: WT-EM-MR-SF-CG (Experimental): Charge: weekly tracking, expert-generated motivational messages, multiple reminders, specific goal feedback, compare to group
  Interventions: Behavioral: Charge
- Arm 17: DT-SM-OR-SS-CS (Experimental): Charge: daily tracking, self-generated motivational messages, one reminder, summary score, compare to self.
  Interventions: Behavioral: Charge
- Arm 18: DT-SM-OR-SS-CG (Experimental): Charge: daily tracking, self-generated motivational messages, one reminder, summary score, compare to group
  Interventions: Behavioral: Charge
- Arm 19: DT-SM-OR-SF-CS (Experimental): Charge: daily tracking, self-generated motivational messages, one reminder, specific goal feedback, compare to self.
  Interventions: Behavioral: Charge
- Arm 20: DT-SM-OR-SF-CG (Experimental): Charge: daily tracking, self-generated motivational messages, one reminder, specific goal feedback, compare to group
  Interventions: Behavioral: Charge
- Arm 21: DT-SM-MR-SS-CS (Experimental): Charge: daily tracking, self-generated motivational messages, multiple reminders, summary score, compare to self
  Interventions: Behavioral: Charge
- Arm 22: DT-SM-MR-SS-CG (Experimental): Charge: daily tracking, self-generated motivational messages, multiple reminders, summary score, compare to group.
  Interventions: Behavioral: Charge
- Arm 23: DT-SM-MR-SF-CS (Experimental): Charge: daily tracking, self-generated motivational messages, multiple reminders, specific goal feedback, compare to self.
  Interventions: Behavioral: Charge
- Arm 24: DT-SM-MR-SF-CG (Experimental): Charge: daily tracking, self-generated motivational messages, multiple reminders, specific goal feedback, compare to group
  Interventions: Behavioral: Charge
- Arm 25: DT-EM-OR-SS-CS (Experimental): Charge: daily tracking, expert-generated motivational messages, one reminder, summary score, compare to self
  Interventions: Behavioral: Charge
- Arm 26: DT-EM-OR-SS-CG (Experimental): Charge: daily tracking, expert-generated motivational messages, one reminder, summary score, compare to group
  Interventions: Behavioral: Charge
- Arm 27: DT-EM-OR-SF-CS (Experimental): Charge: daily tracking, expert-generated motivational messages, one reminder, specific goal feedback, compare to self
  Interventions: Behavioral: Charge
- Arm 28: DT-EM-OR-SF-CG (Experimental): Charge: daily tracking, expert-generated motivational messages, one reminder, specific goal feedback, compare to group
  Interventions: Behavioral: Charge
- Arm 29: DT-EM-MR-SS-CS (Experimental): Charge: daily tracking, expert-generated motivational messages, multiple reminders, summary score, compare to self
  Interventions: Behavioral: Charge
- Arm 30: DT-EM-MR-SS-CG (Experimental): Charge: daily tracking, expert-generated motivational messages, multiple reminders, summary score, compare to group
  Interventions: Behavioral: Charge
- Arm 31: DT-EM-MR-GF-CS (Experimental): Charge: daily tracking, expert-generated motivational messages, multiple reminders, specific goal feedback, compare to self
  Interventions: Behavioral: Charge
- Arm 32: DT-EM-MR-GF-CG (Experimental): Charge: daily tracking, expert-generated motivational messages, multiple reminders, specific goal feedback, compare to group.
  Interventions: Behavioral: Charge

INTERVENTIONS:
Behavioral: Charge — Text messaging-based study to determine effect of different components on weight loss.

SUMMARY:
This study evaluates different versions of a text messaging-based app for weight loss. This study will place participants to 1 of 32 experimental conditions that reflect different texting components and levels. Participants will be randomized to a condition. The investigators will recruit 448 adults into a 6-month weight loss program, with an additional follow-up 6-months after the intervention ends.

DETAILED DESCRIPTION:
Standalone text messaging-based weight loss treatments are scalable and can achieve population reach. However, these interventions are also modular; they can be delivered independently to maximize cost-effectiveness or combined with other approaches (e.g. provider counseling) to maximize outcomes. This study is a 12-month experimental trial among 448 adults with obesity. All participants will receive a core 6-month weight loss texting intervention that includes tailored behavior change goals, interactive self-monitoring, automated feedback, and skills training. Participants will be randomly assigned to 1 of 32 different experimental conditions.

ELIGIBILITY:
Inclusion Criteria:

* males and females aged 18-65 years
* participants have English language proficiency
* participants have a BMI between 25-40 kg/m2
* Participants will own a smartphone
* Participants will be willing to receive multiple text messages daily.

Exclusion Criteria:

* prior or planned bariatric surgery
* psychiatric hospitalization in past 12 months
* pregnancy, nursing, or planned pregnancy
* history of a cardiovascular event
* history of an eating disorder
* history of a condition (e.g., end stage renal disease, cancer, schizophrenia) or use of medications (e.g., lithium, steroids, anti-psychotics) that would affect weight measurement, for which weight loss is contraindicated, or might promote weight change
* current participation in a weight loss trial and/or recent weight loss > 10%
* investigator discretion for safety reasons

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2023-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary G Bennett, PhD, Principal Investigator — Bishop-MacDermott Family Professor of Psychology, Global Health & Medicine
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Collins LM, Baker TB, Mermelstein RJ, Piper ME, Jorenby DE, Smith SS, Christiansen BA, Schlam TR, Cook JW, Fiore MC. The multiphase optimization strategy for engineering effective tobacco use interventions. Ann Behav Med. 2011 Apr;41(2):208-26. doi: 10.1007/s12160-010-9253-x. PMID 21132416
- [Background] Ogden CL, Carroll MD, Flegal KM. Prevalence of obesity in the United States. JAMA. 2014 Jul;312(2):189-90. doi: 10.1001/jama.2014.6228. No abstract available. PMID 25005661
- [Background] Flegal KM, Carroll MD, Kit BK, Ogden CL. Prevalence of obesity and trends in the distribution of body mass index among US adults, 1999-2010. JAMA. 2012 Feb 1;307(5):491-7. doi: 10.1001/jama.2012.39. Epub 2012 Jan 17. PMID 22253363
- [Background] Yang L, Colditz GA. Prevalence of Overweight and Obesity in the United States, 2007-2012. JAMA Intern Med. 2015 Aug;175(8):1412-3. doi: 10.1001/jamainternmed.2015.2405. No abstract available. PMID 26098405
- [Background] Ogden CL, Lamb MM, Carroll MD, Flegal KM. Obesity and socioeconomic status in adults: United States, 2005-2008. NCHS Data Brief. 2010 Dec;(50):1-8. PMID 21211165
- [Background] Rodriguez F, Ferdinand KC. Hypertension in minority populations: new guidelines and emerging concepts. Adv Chronic Kidney Dis. 2015 Mar;22(2):145-53. doi: 10.1053/j.ackd.2014.08.004. PMID 25704352
- [Background] Befort CA, Nazir N, Perri MG. Prevalence of obesity among adults from rural and urban areas of the United States: findings from NHANES (2005-2008). J Rural Health. 2012 Fall;28(4):392-7. doi: 10.1111/j.1748-0361.2012.00411.x. Epub 2012 May 31. PMID 23083085
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. J Am Coll Cardiol. 2014 Jul 1;63(25 Pt B):2985-3023. doi: 10.1016/j.jacc.2013.11.004. Epub 2013 Nov 12. No abstract available. PMID 24239920
- [Background] Mokdad AH, Ford ES, Bowman BA, Dietz WH, Vinicor F, Bales VS, Marks JS. Prevalence of obesity, diabetes, and obesity-related health risk factors, 2001. JAMA. 2003 Jan 1;289(1):76-9. doi: 10.1001/jama.289.1.76. PMID 12503980
- [Background] Finkelstein EA, Brown DS, Wrage LA, Allaire BT, Hoerger TJ. Individual and aggregate years-of-life-lost associated with overweight and obesity. Obesity (Silver Spring). 2010 Feb;18(2):333-9. doi: 10.1038/oby.2009.253. Epub 2009 Aug 13. PMID 19680230
- [Background] Fontaine KR, Redden DT, Wang C, Westfall AO, Allison DB. Years of life lost due to obesity. JAMA. 2003 Jan 8;289(2):187-93. doi: 10.1001/jama.289.2.187. PMID 12517229
- [Background] Han X, Stevens J, Truesdale KP, Bradshaw PT, Kucharska-Newton A, Prizment AE, Platz EA, Joshu CE. Body mass index at early adulthood, subsequent weight change and cancer incidence and mortality. Int J Cancer. 2014 Dec 15;135(12):2900-9. doi: 10.1002/ijc.28930. Epub 2014 May 8. PMID 24771654
- [Background] Osei-Assibey G, Kyrou I, Adi Y, Kumar S, Matyka K. Dietary and lifestyle interventions for weight management in adults from minority ethnic/non-White groups: a systematic review. Obes Rev. 2010 Nov;11(11):769-76. doi: 10.1111/j.1467-789X.2009.00695.x. PMID 20059708
- [Background] Bennett GG, Glasgow RE. The delivery of public health interventions via the Internet: actualizing their potential. Annu Rev Public Health. 2009;30:273-92. doi: 10.1146/annurev.publhealth.031308.100235. PMID 19296777
- [Background] Evans W, Nielsen PE, Szekely DR, Bihm JW, Murray EA, Snider J, Abroms LC. Dose-response effects of the text4baby mobile health program: randomized controlled trial. JMIR Mhealth Uhealth. 2015 Jan 28;3(1):e12. doi: 10.2196/mhealth.3909. PMID 25630361
- [Background] Jordan ET, Ray EM, Johnson P, Evans WD. Text4Baby: using text messaging to improve maternal and newborn health. Nurs Womens Health. 2011 Jun-Jul;15(3):206-12. doi: 10.1111/j.1751-486X.2011.01635.x. No abstract available. PMID 21672170
- [Background] Shapiro JR, Koro T, Doran N, Thompson S, Sallis JF, Calfas K, Patrick K. Text4Diet: a randomized controlled study using text messaging for weight loss behaviors. Prev Med. 2012 Nov;55(5):412-7. doi: 10.1016/j.ypmed.2012.08.011. Epub 2012 Aug 27. PMID 22944150
- [Background] Steinberg DM, Levine EL, Askew S, Foley P, Bennett GG. Daily text messaging for weight control among racial and ethnic minority women: randomized controlled pilot study. J Med Internet Res. 2013 Nov 18;15(11):e244. doi: 10.2196/jmir.2844. PMID 24246427
- [Derived] Bennett GG, Steinberg D, Bolton J, Gallis JA, Treadway C, Askew S, Kay MC, Pollak KI, Turner EL. Optimizing an Obesity Treatment Using the Multiphase Optimization Strategy Framework: Protocol for a Randomized Factorial Trial. JMIR Res Protoc. 2021 Jan 18;10(1):e19506. doi: 10.2196/19506. PMID 33459600

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Those who were eligible and consented to be in the study, prior to randomization.
Groups:
- Experimental: Arm 1: WT-SM-OR-SS-CS: Charge: weekly tracking, self-generated motivational messages, one reminder, summary score, compare to self
- Experimental: Arm 2: WT-SM-OR-SS-CG: Charge: weekly tracking, self-generated motivational messages, one reminder, summary score, compare to group
- Experimental: Arm 3: WT-SM-OR-SF-CS: Charge: weekly tracking, self-generated motivational messages, one reminder, specific goal feedback, compare to self
- Experimental: Arm 4: WT-SM-OR-SF-CG: Charge: weekly tracking, self-generated motivational messages, one reminder, specific goal feedback, compare to group
- Experimental: Arm 5: WT-SM-MR-SS-CS: Charge: weekly tracking, self-generated motivational messages, multiple reminders, summary score, compare to self.
- Experimental: Arm 6: WT-SM-MR-SS-CG: Charge: weekly tracking, self-generated motivational messages, multiple reminders, summary score, compare to group.
- Experimental: Arm 7: WT-SM-MR-SF-CS: Charge: weekly tracking, self-generated motivational messages, multiple reminders, specific feedback, compare to self
- Experimental: Arm 8: WT-SM-MR-SF-CG: Charge: weekly tracking, self-generated motivational messages, multiple reminders, specific feedback, compare to group
- Experimental: Arm 9: WT-EM-OR-SS-CS: Charge: weekly tracking, expert-generated motivational messages, one reminder, summary score, compare to self
- Experimental: Arm 10: WT-EM-OR-SS-CG: Charge: weekly tracking, expert-generated motivational messages, one reminder, summary score, compare to group
- Experimental: Arm 11: WT-EM-OR-SF-CS: Charge: weekly tracking, expert-generated motivational messages, one reminder, specific goal feedback, compare to self
- Experimental: Arm 12: WT-EM-OR-SF-CG: Charge: weekly tracking, expert-generated motivational messages, one reminder, specific goal feedback, compare to group.
- Experimental: Arm 13: WT-EM-MR-SS-CS: Charge: weekly tracking, expert-generated motivational messages, multiple reminders, summary score, compare to self
- Experimental: Arm 14: WT-EM-MR-SS-CG: Charge: weekly tracking, expert-generated motivational messages, multiple reminders,summary score, compare to group
- Experimental: Arm 15: WT-EM-MR-SF-CS: Charge: weekly tracking, expert-generated motivational messages, multiple reminders, specific goal feedback, compare to self
- Experimental: Arm 16: WT-EM-MR-SF-CG: Charge: weekly tracking, expert-generated motivational messages, multiple reminders, specific goal feedback, compare to group
- Experimental: Arm 17: DT-SM-OR-SS-CS: Charge: daily tracking, self-generated motivational messages, one reminder, summary score, compare to self.
- Experimental: Arm 18: DT-SM-OR-SS-CG: Charge: daily tracking, self-generated motivational messages, one reminder, summary score, compare to group
- Experimental: Arm 19: DT-SM-OR-SF-CS: Charge: daily tracking, self-generated motivational messages, one reminder, specific goal feedback, compare to self.
- Experimental: Arm 20: DT-SM-OR-SF-CG: Charge: daily tracking, self-generated motivational messages, one reminder, specific goal feedback, compare to group
- Experimental: Arm 21: DT-SM-MR-SS-CS: Charge: daily tracking, self-generated motivational messages, multiple reminders, summary score, compare to self
- Experimental: Arm 22: DT-SM-MR-SS-CG: Charge: daily tracking, self-generated motivational messages, multiple reminders, summary score, compare to group.
- Experimental: Arm 23: DT-SM-MR-SF-CS: Charge: daily tracking, self-generated motivational messages, multiple reminders, specific goal feedback, compare to self.
- Experimental: Arm 24: DT-SM-MR-SF-CG: Charge: daily tracking, self-generated motivational messages, multiple reminders, specific goal feedback, compare to group
- Experimental: Arm 25: DT-EM-OR-SS-CS: Charge: daily tracking, expert-generated motivational messages, one reminder, summary score, compare to self
- Experimental: Arm 26: DT-EM-OR-SS-CG: Charge: daily tracking, expert-generated motivational messages, one reminder, summary score, compare to group
- Experimental: Arm 27: DT-EM-OR-SF-CS: Charge: daily tracking, expert-generated motivational messages, one reminder, specific goal feedback, compare to self
- Experimental: Arm 28: DT-EM-OR-SF-CG: Charge: daily tracking, expert-generated motivational messages, one reminder, specific goal feedback, compare to group
- Experimental: Arm 29: DT-EM-MR-SS-CS: Charge: daily tracking, expert-generated motivational messages, multiple reminders, summary score, compare to self
- Experimental: Arm 30: DT-EM-MR-SS-CG: Charge: daily tracking, expert-generated motivational messages, multiple reminders, summary score, compare to group
- Experimental: Arm 31: DT-EM-MR-GF-CS: Charge: daily tracking, expert-generated motivational messages, multiple reminders, specific goal feedback, compare to self
- Experimental: Arm 32: DT-EM-MR-GF-CG: Charge: daily tracking, expert-generated motivational messages, multiple reminders, specific goal feedback, compare to group.
Period: Overall Study
Arm/Group | Experimental: Arm 1: WT-SM-OR-SS-CS | Experimental: Arm 2: WT-SM-OR-SS-CG | Experimental: Arm 3: WT-SM-OR-SF-CS | Experimental: Arm 4: WT-SM-OR-SF-CG | Experimental: Arm 5: WT-SM-MR-SS-CS | Experimental: Arm 6: WT-SM-MR-SS-CG | Experimental: Arm 7: WT-SM-MR-SF-CS | Experimental: Arm 8: WT-SM-MR-SF-CG | Experimental: Arm 9: WT-EM-OR-SS-CS | Experimental: Arm 10: WT-EM-OR-SS-CG | Experimental: Arm 11: WT-EM-OR-SF-CS | Experimental: Arm 12: WT-EM-OR-SF-CG | Experimental: Arm 13: WT-EM-MR-SS-CS | Experimental: Arm 14: WT-EM-MR-SS-CG | Experimental: Arm 15: WT-EM-MR-SF-CS | Experimental: Arm 16: WT-EM-MR-SF-CG | Experimental: Arm 17: DT-SM-OR-SS-CS | Experimental: Arm 18: DT-SM-OR-SS-CG | Experimental: Arm 19: DT-SM-OR-SF-CS | Experimental: Arm 20: DT-SM-OR-SF-CG | Experimental: Arm 21: DT-SM-MR-SS-CS | Experimental: Arm 22: DT-SM-MR-SS-CG | Experimental: Arm 23: DT-SM-MR-SF-CS | Experimental: Arm 24: DT-SM-MR-SF-CG | Experimental: Arm 25: DT-EM-OR-SS-CS | Experimental: Arm 26: DT-EM-OR-SS-CG | Experimental: Arm 27: DT-EM-OR-SF-CS | Experimental: Arm 28: DT-EM-OR-SF-CG | Experimental: Arm 29: DT-EM-MR-SS-CS | Experimental: Arm 30: DT-EM-MR-SS-CG | Experimental: Arm 31: DT-EM-MR-GF-CS | Experimental: Arm 32: DT-EM-MR-GF-CG
Started | 17 | 16 | 17 | 17 | 16 | 15 | 17 | 17 | 18 | 17 | 18 | 16 | 16 | 15 | 18 | 16 | 18 | 16 | 15 | 17 | 18 | 16 | 15 | 17 | 18 | 17 | 17 | 17 | 16 | 15 | 19 | 17
Completed | 11 | 12 | 10 | 14 | 11 | 11 | 13 | 13 | 13 | 13 | 9 | 13 | 14 | 10 | 12 | 13 | 14 | 12 | 11 | 11 | 13 | 10 | 9 | 12 | 12 | 14 | 13 | 15 | 12 | 13 | 13 | 12
Not Completed | 6 | 4 | 7 | 3 | 5 | 4 | 4 | 4 | 5 | 4 | 9 | 3 | 2 | 5 | 6 | 3 | 4 | 4 | 4 | 6 | 5 | 6 | 6 | 5 | 6 | 3 | 4 | 2 | 4 | 2 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Arm 1: WT-SM-OR-SS-CS | Experimental: Arm 2: WT-SM-OR-SS-CG | Experimental: Arm 3: WT-SM-OR-SF-CS | Experimental: Arm 4: WT-SM-OR-SF-CG | Experimental: Arm 5: WT-SM-MR-SS-CS | Experimental: Arm 6: WT-SM-MR-SS-CG | Experimental: Arm 7: WT-SM-MR-SF-CS | Experimental: Arm 8: WT-SM-MR-SF-CG | Experimental: Arm 9: WT-EM-OR-SS-CS | Experimental: Arm 10: WT-EM-OR-SS-CG | Experimental: Arm 11: WT-EM-OR-SF-CS | Experimental: Arm 12: WT-EM-OR-SF-CG | Experimental: Arm 13: WT-EM-MR-SS-CS | Experimental: Arm 14: WT-EM-MR-SS-CG | Experimental: Arm 15: WT-EM-MR-SF-CS | Experimental: Arm 16: WT-EM-MR-SF-CG | Experimental: Arm 17: DT-SM-OR-SS-CS | Experimental: Arm 18: DT-SM-OR-SS-CG | Experimental: Arm 19: DT-SM-OR-SF-CS | Experimental: Arm 20: DT-SM-OR-SF-CG | Experimental: Arm 21: DT-SM-MR-SS-CS | Experimental: Arm 22: DT-SM-MR-SS-CG | Experimental: Arm 23: DT-SM-MR-SF-CS | Experimental: Arm 24: DT-SM-MR-SF-CG | Experimental: Arm 25: DT-EM-OR-SS-CS | Experimental: Arm 26: DT-EM-OR-SS-CG | Experimental: Arm 27: DT-EM-OR-SF-CS | Experimental: Arm 28: DT-EM-OR-SF-CG | Experimental: Arm 29: DT-EM-MR-SS-CS | Experimental: Arm 30: DT-EM-MR-SS-CG | Experimental: Arm 31: DT-EM-MR-GF-CS | Experimental: Arm 32: DT-EM-MR-GF-CG | Total
Number analyzed (Participants) | 17 | 16 | 17 | 17 | 16 | 15 | 17 | 17 | 18 | 17 | 18 | 16 | 16 | 15 | 18 | 16 | 18 | 16 | 15 | 17 | 18 | 16 | 15 | 17 | 18 | 17 | 17 | 17 | 16 | 15 | 19 | 17 | 534
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 17 | 17 | 16 | 15 | 17 | 17 | 18 | 17 | 18 | 16 | 16 | 15 | 17 | 16 | 18 | 16 | 15 | 17 | 18 | 16 | 14 | 17 | 18 | 16 | 17 | 17 | 16 | 15 | 19 | 16 | 530
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (8.3) | 39.5 (12.3) | 46.8 (10.7) | 44.4 (12.6) | 39.4 (10.5) | 46.5 (11.8) | 40.2 (14.9) | 41.2 (11.8) | 37.2 (8.7) | 43.0 (12.8) | 42.8 (13.9) | 41.0 (11.6) | 45.4 (13.7) | 45.2 (12.9) | 41.2 (13.3) | 40.6 (11.6) | 42.6 (13.2) | 44.9 (12.4) | 42.0 (10.9) | 41.2 (11.7) | 42.6 (12.4) | 37.9 (7.8) | 43.2 (14.0) | 34.4 (5.4) | 33.4 (5.5) | 36.3 (6.4) | 33.4 (6.2) | 32.5 (6.1) | 36.6 (7.1) | 34.3 (3.7) | 32.0 (4.8) | 34.6 (7.8) | 33.9 (6.1)
Sex/Gender, Customized [Count of Participants; unit: Participants] — We asked participants to identify as male, male or Other (self described)
  Participants
    Gender - Self Described: Other (self described as genderqueer or nonbinary) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
    Gender - Self Described: Male | 5 | 5 | 4 | 4 | 4 | 4 | 5 | 5 | 5 | 5 | 5 | 4 | 4 | 4 | 6 | 4 | 5 | 4 | 4 | 4 | 5 | 5 | 4 | 4 | 5 | 4 | 5 | 5 | 4 | 4 | 5 | 5 | 145
    Gender - Self Described: Female | 12 | 11 | 13 | 13 | 12 | 11 | 12 | 12 | 13 | 12 | 12 | 12 | 12 | 11 | 12 | 12 | 13 | 12 | 11 | 13 | 12 | 11 | 11 | 13 | 13 | 13 | 12 | 12 | 12 | 11 | 13 | 12 | 386
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Non-Hispanic Black | 1 | 0 | 2 | 4 | 3 | 4 | 2 | 2 | 5 | 4 | 2 | 2 | 2 | 3 | 3 | 4 | 1 | 1 | 3 | 3 | 3 | 3 | 5 | 2 | 0 | 2 | 1 | 2 | 4 | 0 | 1 | 3 | 77
  Race/Ethnicity: Non-Hispanic White | 11 | 14 | 15 | 12 | 10 | 10 | 10 | 13 | 11 | 11 | 15 | 11 | 12 | 10 | 11 | 11 | 13 | 15 | 11 | 10 | 13 | 12 | 10 | 14 | 13 | 14 | 12 | 13 | 9 | 14 | 18 | 13 | 391
  Race/Ethnicity: Hispanic (all races) | 2 | 1 | 0 | 0 | 3 | 0 | 1 | 1 | 2 | 0 | 0 | 3 | 2 | 1 | 3 | 1 | 3 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 3 | 0 | 0 | 1 | 36
  Race/Ethnicity: Non-Hispanic Other | 3 | 1 | 0 | 1 | 0 | 1 | 4 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 3 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 30
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 17 | 17 | 16 | 15 | 17 | 17 | 18 | 17 | 18 | 16 | 16 | 15 | 18 | 16 | 18 | 16 | 15 | 17 | 18 | 16 | 15 | 17 | 18 | 17 | 17 | 17 | 16 | 15 | 19 | 17 | 534
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.1 (6) | 33.2 (5.9) | 30.6 (2.8) | 32.7 (6.2) | 34.9 (7.2) | 33.9 (7.2) | 32.4 (7.5) | 35.9 (7.3) | 36.9 (8.3) | 32.1 (5.2) | 34.4 (7.2) | 33.7 (4.4) | 35.8 (5.4) | 32.5 (5.7) | 36.7 (6.4) | 32.8 (4.9) | 32.1 (4.6) | 34.9 (6.1) | 32.9 (5.6) | 32.8 (4.6) | 33.6 (5.5) | 36.2 (7.9) | 33.9 (6.6) | 34.4 (5.4) | 33.4 (5.5) | 36.3 (6.4) | 33.4 (6.2) | 32.5 (6.1) | 36.6 (7.1) | 34.3 (3.7) | 32.0 (4.8) | 34.6 (7.7) | 33.9 (6.1)
Personal income [Count of Participants; unit: Participants]
  Missing | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 20
  Less than $25,000 | 6 | 2 | 2 | 1 | 4 | 2 | 6 | 4 | 5 | 0 | 1 | 4 | 3 | 4 | 5 | 4 | 3 | 2 | 1 | 3 | 3 | 2 | 1 | 7 | 4 | 3 | 8 | 0 | 1 | 4 | 3 | 2 | 100
  $25,000 through $49,999 | 2 | 6 | 4 | 4 | 7 | 6 | 3 | 3 | 8 | 6 | 6 | 4 | 5 | 5 | 3 | 3 | 5 | 5 | 1 | 2 | 4 | 2 | 5 | 2 | 4 | 2 | 2 | 4 | 8 | 3 | 6 | 5 | 135
  $50,000 and greater | 9 | 7 | 11 | 10 | 5 | 7 | 8 | 10 | 4 | 10 | 11 | 7 | 6 | 6 | 9 | 9 | 10 | 9 | 10 | 11 | 10 | 12 | 8 | 8 | 9 | 10 | 7 | 12 | 7 | 7 | 10 | 10 | 279

OUTCOME MEASURES:

1. Primary Outcome: Average Weight Change
Description: Mean change in weight in kg (6 months post-randomization- baseline weight)
Time Frame: baseline, 6 months
Population: The primary outcome was 6-month change in weight (kg), measured at each in-person visit.
Measure: Mean (Standard Deviation); unit: Weight in kg
Arm/Group | Experimental: Arm 1: WT-SM-OR-SS-CS | Experimental: Arm 2: WT-SM-OR-SS-CG | Experimental: Arm 3: WT-SM-OR-SF-CS | Experimental: Arm 4: WT-SM-OR-SF-CG | Experimental: Arm 5: WT-SM-MR-SS-CS | Experimental: Arm 6: WT-SM-MR-SS-CG | Experimental: Arm 7: WT-SM-MR-SF-CS | Experimental: Arm 8: WT-SM-MR-SF-CG | Experimental: Arm 9: WT-EM-OR-SS-CS | Experimental: Arm 10: WT-EM-OR-SS-CG | Experimental: Arm 11: WT-EM-OR-SF-CS | Experimental: Arm 12: WT-EM-OR-SF-CG | Experimental: Arm 13: WT-EM-MR-SS-CS | Experimental: Arm 14: WT-EM-MR-SS-CG | Experimental: Arm 15: WT-EM-MR-SF-CS | Experimental: Arm 16: WT-EM-MR-SF-CG | Experimental: Arm 17: DT-SM-OR-SS-CS | Experimental: Arm 18: DT-SM-OR-SS-CG | Experimental: Arm 19: DT-SM-OR-SF-CS | Experimental: Arm 20: DT-SM-OR-SF-CG | Experimental: Arm 21: DT-SM-MR-SS-CS | Experimental: Arm 22: DT-SM-MR-SS-CG | Experimental: Arm 23: DT-SM-MR-SF-CS | Experimental: Arm 24: DT-SM-MR-SF-CG | Experimental: Arm 25: DT-EM-OR-SS-CS | Experimental: Arm 26: DT-EM-OR-SS-CG | Experimental: Arm 27: DT-EM-OR-SF-CS | Experimental: Arm 28: DT-EM-OR-SF-CG | Experimental: Arm 29: DT-EM-MR-SS-CS | Experimental: Arm 30: DT-EM-MR-SS-CG | Experimental: Arm 31: DT-EM-MR-GF-CS | Experimental: Arm 32: DT-EM-MR-GF-CG
Number analyzed (Participants) | 11 | 12 | 10 | 14 | 11 | 11 | 13 | 13 | 13 | 13 | 9 | 13 | 14 | 10 | 12 | 13 | 14 | 12 | 11 | 11 | 13 | 10 | 9 | 12 | 12 | 14 | 13 | 15 | 12 | 13 | 13 | 12
Weight in kg | 0.1 (3.3) | -0.4 (2.7) | -3.4 (4.3) | -0.8 (4.8) | -3.3 (8.1) | -1.3 (5.8) | -0.9 (5.6) | -2.3 (5.6) | -2.9 (3.8) | -0.7 (2.3) | -1.0 (3.6) | -3.0 (5.8) | -2.9 (6.5) | -1.5 (2.3) | -2.1 (7.2) | -2.5 (2.8) | -3.1 (4.3) | -4.5 (5.9) | -2.8 (2.7) | -1.9 (4.6) | -1.5 (3.0) | -0.3 (4.1) | -0.5 (2.2) | -1.0 (5.9) | -2.7 (6.3) | -3.3 (6.2) | -2.4 (5.5) | -1.8 (3.3) | -3.5 (6.2) | -2.8 (6.4) | 0.2 (3.6) | -1.0 (6.5)

2. Secondary Outcome: Change in Diet
Description: To experimentally determine the effects of text messaging components and levels on change in dietary intake using The Rapid Eating Assessment for Participants - Shortened version (REAP-S). The range of score is 13 to 39, where a higher score indicates more healthy dietary intake.
Time Frame: baseline, 6 months
Population: Average change in REAP-S score (6-months - baseline).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: WT-SM-OR-SS-CS | Arm 2: WT-SM-OR-SS-CG | Arm 3: WT-SM-OR-SF-CS | Arm 4: WT-SM-OR-SF-CG | Arm 5: WT-SM-MR-SS-CS | Arm 6: WT-SM-MR-SS-CG | Arm 7: WT-SM-MR-SF-CS | Arm 8: WT-SM-MR-SF-CG | Arm 9: WT-EM-OR-SS-CS | Arm 10: WT-EM-OR-SS-CG | Arm 11: WT-EM-OR-SF-CS | Arm 12: WT-EM-OR-SF-CG | Arm 13: WT-EM-MR-SS-CS | Arm 14: WT-EM-MR-SS-CG | Arm 15: WT-EM-MR-SF-CS | Arm 16: WT-EM-MR-SF-CG | Arm 17: DT-SM-OR-SS-CS | Arm 18: DT-SM-OR-SS-CG | Arm 19: DT-SM-OR-SF-CS | Arm 20: DT-SM-OR-SF-CG | Arm 21: DT-SM-MR-SS-CS | Arm 22: DT-SM-MR-SS-CG | Arm 23: DT-SM-MR-SF-CS | Arm 24: DT-SM-MR-SF-CG | Arm 25: DT-EM-OR-SS-CS | Arm 26: DT-EM-OR-SS-CG | Arm 27: DT-EM-OR-SF-CS | Arm 28: DT-EM-OR-SF-CG | Arm 29: DT-EM-MR-SS-CS | Arm 30: DT-EM-MR-SS-CG | Arm 31: DT-EM-MR-GF-CS | Arm 32: DT-EM-MR-GF-CG
Number analyzed (Participants) | 12 | 14 | 11 | 15 | 12 | 12 | 13 | 13 | 16 | 14 | 8 | 14 | 15 | 10 | 15 | 13 | 15 | 13 | 13 | 13 | 16 | 12 | 10 | 13 | 12 | 15 | 14 | 15 | 15 | 14 | 14 | 13
score on a scale | 0.8 (4) | 2 (5) | 4.4 (3.1) | 1.2 (3.8) | 3.8 (5.8) | 2.6 (3.4) | 1.8 (3.5) | 1.8 (3.9) | 1.8 (3.5) | 2 (2.9) | 2.4 (3.2) | 2.2 (3.6) | 2.7 (3.3) | 2.9 (2.7) | 3.3 (4.7) | 1.5 (2.3) | 2.4 (3.1) | 3.7 (4.8) | 1.4 (2.5) | 0.4 (3.2) | 2.8 (3.6) | 1.1 (4.6) | 2.5 (2.9) | 1.5 (2.5) | 1.1 (4.6) | 3.8 (3.1) | 2.9 (4.1) | 1.2 (3.4) | 1.9 (2.5) | 1.6 (2.7) | 0.9 (4.0) | 3.7 (4.7)

3. Secondary Outcome: Average Change in Physical Activity
Description: To experimentally determine the effects of text messaging components and levels on change in weekly minutes of physical activity based on the WHO Global Physical Activity Questionnaire version 2 (GPAC 2). The range of scores is 0 minutes/week to 10,080 minutes/week (maximum number of minutes in a week).
Time Frame: baseline, 6 months
Population: Average difference of GPAC 2 scores at 6 months as compared to baseline
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | Experimental: Arm 1: WT-SM-OR-SS-CS | Experimental: Arm 2: WT-SM-OR-SS-CG | Experimental: Arm 3: WT-SM-OR-SF-CS | Experimental: Arm 4: WT-SM-OR-SF-CG | Experimental: Arm 5: WT-SM-MR-SS-CS | Experimental: Arm 6: WT-SM-MR-SS-CG | Experimental: Arm 7: WT-SM-MR-SF-CS | Experimental: Arm 8: WT-SM-MR-SF-CG | Experimental: Arm 9: WT-EM-OR-SS-CS | Experimental: Arm 10: WT-EM-OR-SS-CG | Experimental: Arm 11: WT-EM-OR-SF-CS | Experimental: Arm 12: WT-EM-OR-SF-CG | Experimental: Arm 13: WT-EM-MR-SS-CS | Experimental: Arm 14: WT-EM-MR-SS-CG | Experimental: Arm 15: WT-EM-MR-SF-CS | Experimental: Arm 16: WT-EM-MR-SF-CG | Experimental: Arm 17: DT-SM-OR-SS-CS | Experimental: Arm 18: DT-SM-OR-SS-CG | Experimental: Arm 19: DT-SM-OR-SF-CS | Experimental: Arm 20: DT-SM-OR-SF-CG | Experimental: Arm 21: DT-SM-MR-SS-CS | Experimental: Arm 22: DT-SM-MR-SS-CG | Experimental: Arm 23: DT-SM-MR-SF-CS | Experimental: Arm 24: DT-SM-MR-SF-CG | Experimental: Arm 25: DT-EM-OR-SS-CS | Experimental: Arm 26: DT-EM-OR-SS-CG | Experimental: Arm 27: DT-EM-OR-SF-CS | Experimental: Arm 28: DT-EM-OR-SF-CG | Experimental: Arm 29: DT-EM-MR-SS-CS | Experimental: Arm 30: DT-EM-MR-SS-CG | Experimental: Arm 31: DT-EM-MR-GF-CS | Experimental: Arm 32: DT-EM-MR-GF-CG
Number analyzed (Participants) | 9 | 13 | 11 | 13 | 11 | 8 | 10 | 12 | 13 | 12 | 8 | 11 | 13 | 7 | 14 | 11 | 15 | 13 | 11 | 11 | 13 | 12 | 8 | 12 | 11 | 15 | 13 | 15 | 13 | 11 | 13 | 11
minutes per week | 202.2 (718.6) | 103.8 (208.5) | 256.8 (762.0) | 335.6 (449.9) | 88.6 (138.2) | 241.5 (684.8) | 390.6 (859.0) | 202.9 (385.5) | 106.9 (285.8) | 159.2 (381.2) | 143.1 (413.5) | 319.1 (620.3) | 81.2 (754.5) | 390.0 (732.4) | 41.1 (208.1) | -26.4 (274.2) | -76.5 (382.6) | 70.0 (548.8) | 48.2 (264.0) | -362.7 (2225.4) | 45.0 (154.1) | 75.0 (171.6) | -54.4 (525.8) | 95.9 (325.8) | 197.7 (401.9) | 201.3 (646.4) | 105.8 (419.4) | -21.3 (418.1) | -76.9 (272.2) | 408.2 (652.0) | 505.5 (1167.1) | 48.6 (302.4)

ADVERSE EVENTS:
Time Frame: 1 year, 5 months
Description: We used clinicaltrials.gov definitions and collected adverse event information at study visits.
Arm/Group | Experimental: Arm 1: WT-SM-OR-SS-CS | Experimental: Arm 2: WT-SM-OR-SS-CG | Experimental: Arm 3: WT-SM-OR-SF-CS | Experimental: Arm 4: WT-SM-OR-SF-CG | Experimental: Arm 5: WT-SM-MR-SS-CS | Experimental: Arm 6: WT-SM-MR-SS-CG | Experimental: Arm 7: WT-SM-MR-SF-CS | Experimental: Arm 8: WT-SM-MR-SF-CG | Experimental: Arm 9: WT-EM-OR-SS-CS | Experimental: Arm 10: WT-EM-OR-SS-CG | Experimental: Arm 11: WT-EM-OR-SF-CS | Experimental: Arm 12: WT-EM-OR-SF-CG | Experimental: Arm 13: WT-EM-MR-SS-CS | Experimental: Arm 14: WT-EM-MR-SS-CG | Experimental: Arm 15: WT-EM-MR-SF-CS | Experimental: Arm 16: WT-EM-MR-SF-CG | Experimental: Arm 17: DT-SM-OR-SS-CS | Experimental: Arm 18: DT-SM-OR-SS-CG | Experimental: Arm 19: DT-SM-OR-SF-CS | Experimental: Arm 20: DT-SM-OR-SF-CG | Experimental: Arm 21: DT-SM-MR-SS-CS | Experimental: Arm 22: DT-SM-MR-SS-CG | Experimental: Arm 23: DT-SM-MR-SF-CS | Experimental: Arm 24: DT-SM-MR-SF-CG | Experimental: Arm 25: DT-EM-OR-SS-CS | Experimental: Arm 26: DT-EM-OR-SS-CG | Experimental: Arm 27: DT-EM-OR-SF-CS | Experimental: Arm 28: DT-EM-OR-SF-CG | Experimental: Arm 29: DT-EM-MR-SS-CS | Experimental: Arm 30: DT-EM-MR-SS-CG | Experimental: Arm 31: DT-EM-MR-GF-CS | Experimental: Arm 32: DT-EM-MR-GF-CG
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16 | 0/17 | 0/17 | 0/16 | 0/15 | 0/17 | 0/17 | 0/18 | 0/17 | 0/18 | 0/16 | 0/16 | 0/15 | 0/18 | 0/16 | 0/18 | 0/16 | 0/15 | 0/17 | 0/18 | 0/16 | 0/15 | 0/17 | 0/18 | 0/17 | 0/17 | 0/17 | 0/16 | 0/15 | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/17 | 0/17 | 0/16 | 0/15 | 0/17 | 0/17 | 0/18 | 0/17 | 0/18 | 0/16 | 0/16 | 0/15 | 0/18 | 0/16 | 0/18 | 0/16 | 0/15 | 0/17 | 0/18 | 0/16 | 0/15 | 0/17 | 0/18 | 0/17 | 0/17 | 0/17 | 0/16 | 0/15 | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16 | 0/17 | 0/17 | 0/16 | 0/15 | 0/17 | 0/17 | 0/18 | 0/17 | 0/18 | 0/16 | 0/16 | 0/15 | 1/18 | 0/16 | 0/18 | 0/16 | 0/15 | 0/17 | 0/18 | 0/16 | 0/15 | 0/17 | 0/18 | 0/17 | 0/17 | 0/17 | 0/16 | 0/15 | 0/19 | 0/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Arm 1: WT-SM-OR-SS-CS (N=17) | Experimental: Arm 2: WT-SM-OR-SS-CG (N=16) | Experimental: Arm 3: WT-SM-OR-SF-CS (N=17) | Experimental: Arm 4: WT-SM-OR-SF-CG (N=17) | Experimental: Arm 5: WT-SM-MR-SS-CS (N=16) | Experimental: Arm 6: WT-SM-MR-SS-CG (N=15) | Experimental: Arm 7: WT-SM-MR-SF-CS (N=17) | Experimental: Arm 8: WT-SM-MR-SF-CG (N=17) | Experimental: Arm 9: WT-EM-OR-SS-CS (N=18) | Experimental: Arm 10: WT-EM-OR-SS-CG (N=17) | Experimental: Arm 11: WT-EM-OR-SF-CS (N=18) | Experimental: Arm 12: WT-EM-OR-SF-CG (N=16) | Experimental: Arm 13: WT-EM-MR-SS-CS (N=16) | Experimental: Arm 14: WT-EM-MR-SS-CG (N=15) | Experimental: Arm 15: WT-EM-MR-SF-CS (N=18) | Experimental: Arm 16: WT-EM-MR-SF-CG (N=16) | Experimental: Arm 17: DT-SM-OR-SS-CS (N=18) | Experimental: Arm 18: DT-SM-OR-SS-CG (N=16) | Experimental: Arm 19: DT-SM-OR-SF-CS (N=15) | Experimental: Arm 20: DT-SM-OR-SF-CG (N=17) | Experimental: Arm 21: DT-SM-MR-SS-CS (N=18) | Experimental: Arm 22: DT-SM-MR-SS-CG (N=16) | Experimental: Arm 23: DT-SM-MR-SF-CS (N=15) | Experimental: Arm 24: DT-SM-MR-SF-CG (N=17) | Experimental: Arm 25: DT-EM-OR-SS-CS (N=18) | Experimental: Arm 26: DT-EM-OR-SS-CG (N=17) | Experimental: Arm 27: DT-EM-OR-SF-CS (N=17) | Experimental: Arm 28: DT-EM-OR-SF-CG (N=17) | Experimental: Arm 29: DT-EM-MR-SS-CS (N=16) | Experimental: Arm 30: DT-EM-MR-SS-CG (N=15) | Experimental: Arm 31: DT-EM-MR-GF-CS (N=19) | Experimental: Arm 32: DT-EM-MR-GF-CG (N=17)
Low blood sugar (hypoglycemia) (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/40/NCT03254940/Prot_SAP_ICF_000.pdf